CLINICAL TRIAL: NCT07242144
Title: A Prospective Observational Study on the Effect of Changes in Endotracheal Tube Cuff Pressure on Postoperative Pharyngolaryngeal Complications in Patients Undergoing Robot-Assisted Radical Prostatectomy
Brief Title: Effect of Changes in Endotracheal Tube Cuff Pressure on Postoperative Pharyngolaryngeal Complications in Robotic Surgery
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nursen Karaca, Medical Doctor, Ege University
Other Study IDs: EUTF 23-7/3
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Robot-Assisted Radical Prostatectomy; Prostatic Neoplasms
Keywords: Endotracheal tube cuff pressure; postoperative pharyngolaryngeal complications; Robot-Assisted Radical Prostatectomy; pneumoperitoneum; steep Trendelenburg position
MeSH Terms: conditions — Prostatic Neoplasms; Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot-Assisted Radical Prostatectomy (RALP): Patients undergoing robot-assisted laparoscopic radical prostatectomy under general anesthesia with a steep Trendelenburg position and pneumoperitoneum
  Interventions: Other: Continuous Monitoring of Endotracheal Tube Cuff Pressure
- Open Radical Prostatectomy (ORP): Patients undergoing open radical prostatectomy under general anesthesia without Trendelenburg position or pneumoperitoneum.
  Interventions: Other: Continuous Monitoring of Endotracheal Tube Cuff Pressure

INTERVENTIONS:
Other: Continuous Monitoring of Endotracheal Tube Cuff Pressure — Continuous intraoperative measurement of endotracheal tube cuff pressure using a manometer at predefined intraoperative time points (after intubation, after pneumoperitoneum, after Trendelenburg positioning, and every 15 minutes thereafter).

SUMMARY:
The goal of this observational study is to evaluate how changes in endotracheal tube (ETT) cuff pressure during robot-assisted radical prostatectomy (RARP) affect postoperative throat-related symptoms. The main question the study aims to answer is: Do pneumoperitoneum and the steep Trendelenburg position used in robotic prostate surgery increase ETT cuff pressure and lead to a higher incidence of postoperative pharyngolaryngeal complications such as sore throat, hoarseness, or dysphagia? This study includes 50 male patients undergoing elective radical prostatectomy under general anesthesia, with 25 patients in the open surgery group and 25 in the robotic-assisted group. The ETT cuff pressure is initially adjusted to the lowest level that prevents air leakage (20-35 cmH#O) and is continuously monitored throughout surgery. Measurements are recorded at specific intraoperative time points related to pneumoperitoneum and positioning. After surgery, patients are evaluated at 2 and 24 hours postoperatively for throat-related symptoms such as sore throat, hoarseness, dysphagia, and cough. The results are expected to clarify whether intraoperative factors unique to robotic surgery contribute to increased cuff pressure and postoperative discomfort, emphasizing the importance of continuous cuff pressure monitoring and timely adjustment for patient safety.

DETAILED DESCRIPTION:
Endotracheal tube (ETT) cuff pressure management is critical in maintaining airway safety during general anesthesia. Excessive cuff pressure may cause mucosal ischemia and postoperative complications such as sore throat, hoarseness, and dysphagia, while insufficient pressure can lead to air leakage and aspiration risk. During robot-assisted laparoscopic radical prostatectomy (RARP), patients are placed in a steep Trendelenburg position with pneumoperitoneum, which may significantly affect airway mechanics and ETT cuff pressure due to increased intrathoracic and airway pressures. This observational study aims to investigate how intraoperative factors unique to robotic surgery-particularly pneumoperitoneum and Trendelenburg positioning-affect ETT cuff pressure and postoperative pharyngolaryngeal outcomes. Fifty adult male patients scheduled for elective radical prostatectomy under general anesthesia are included. Twenty-five undergo open surgery, and twenty-five undergo robotic-assisted surgery. After intubation, the ETT cuff is inflated to the minimal occlusive volume (20-35 cmH#O) and monitored continuously throughout the procedure. Cuff pressure measurements are obtained at defined intraoperative time points, including after pneumoperitoneum, following positioning, and periodically during surgery. Postoperative evaluation includes structured interviews at 2 and 24 hours after extubation to document throat-related symptoms such as sore throat, hoarseness, dysphagia, and cough. The study seeks to provide practical evidence on whether robotic surgical positioning and pneumoperitoneum contribute to elevated cuff pressure and subsequent airway discomfort. These findings may highlight the need for continuous cuff pressure monitoring and adjustment during robot-assisted procedures to improve patient safety and postoperative comfort.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 40 to 80 years

  * Classified as American Society of Anesthesiologists (ASA) physical status I-II
  * Scheduled for elective robot-assisted laparoscopic radical prostatectomy (RALP) or open radical prostatectomy under general anesthesia
  * Able to understand the study procedure and provide written informed consent

Exclusion Criteria:

* • Emergency surgery

  * Upper or lower respiratory tract infection within 10 days before surgery
  * ASA physical status > III
  * Obstructed or kinked intraoperative endotracheal tube
  * Risk of aspiration (e.g., gastroesophageal reflux, full stomach)
  * Preoperative sore throat or existing pharyngolaryngeal symptoms
  * Body mass index (BMI) > 35 kg/m²

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of male patients aged 40 to 80 years who underwent elective robot-assisted laparoscopic radical prostatectomy (RALP) or open radical prostatectomy under general anesthesia at Ege University Faculty of Medicine Hospital. All participants were classified as American Society of Anesthesiologists (ASA) physical status I-II and provided written informed consent prior to inclusion
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Pharyngolaryngeal Complications | Within 24 hours postoperatively
  Presence of cough assessed at 2 and 24 hours after extubation.
Change in Endotracheal Tube Cuff Pressure During Surgery | Intraoperative period (from induction to end of surgery)]
  Endotracheal tube cuff pressure will be continuously monitored from intubation (T1) through various intraoperative stages, including pneumoperitoneum, Trendelenburg positioning, and desufflation

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Medical Faculty Department of Anesthesiology and Reanimation, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single center observational study with a small patient population and institutional confidentiality restrictions.

REFERENCES:
- [Background] Zhu G, Wang X, Cao X, Yang C, Wang B, Ang Y, Duan M. The effect of different endotracheal tube cuff pressure monitoring systems on postoperative sore throat in patients undergoing tracheal intubation: a randomized clinical trial. BMC Anesthesiol. 2024 Mar 25;24(1):115. doi: 10.1186/s12871-024-02499-5. PMID 38528475
- [Background] Liu J, Zhang X, Gong W, Li S, Wang F, Fu S, Zhang M, Hang Y. Correlations between controlled endotracheal tube cuff pressure and postprocedural complications: a multicenter study. Anesth Analg. 2010 Nov;111(5):1133-7. doi: 10.1213/ANE.0b013e3181f2ecc7. Epub 2010 Aug 24. PMID 20736432
- [Background] Phong SV, Koh LK. Anaesthesia for robotic-assisted radical prostatectomy: considerations for laparoscopy in the Trendelenburg position. Anaesth Intensive Care. 2007 Apr;35(2):281-5. doi: 10.1177/0310057X0703500221. PMID 17444322
- [Background] Tsunoda N, Asai T, Okuda Y. Tracheal tube cuff pressure during anesthesia for robotic-assisted laparoscopic prostatectomy and the efficacy of an automatic cuff pressure controller (SmartCuff): observational studies of 1-sample paired data. J Anesth. 2023 Apr;37(2):234-241. doi: 10.1007/s00540-022-03151-7. Epub 2022 Dec 16. PMID 36525125